CLINICAL TRIAL: NCT05583760
Title: Stabilometric and Baropodometric Evaluation of Osteopathic Scaphoid Tug Manipulation
Brief Title: Stabilometric and Baropodometric Evaluation After Osteopathic Scaphoid Tug Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, SERGIO MONTERO NAVARRO, Principal Investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEEI22/322
Record Dates: First submitted 2022-10-10; First posted 2022-10-18 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Manipulation; Osteopathic

STUDY DESIGN:
Who Masked: Participant
Masking Description: SINGLE BLIND (PARTICIPANT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Osteopathic manipulation TUG for scaphoid bone (Experimental)
  Interventions: Procedure: Experimental: Osteopathic manipulation TUG for scaphoid bone
- Sham group: Sham osteopathic manipulation TUG for scaphoid bone (Sham Comparator)
  Interventions: Procedure: Sham group: Sham osteopathic manipulation TUG for scaphoid bone

INTERVENTIONS:
Procedure: Experimental: Osteopathic manipulation TUG for scaphoid bone — The sequence of execution of the scaphoid TUG technique shall be applied as follows. Patient in the supine position. The inner hand of the intervener makes contact with the pisiform through the hypothenar eminence and ulnar border of the hand over the scaphoid tubercle, the outer hand reinforces the contact. The thumbs are directed to the sole of the patient's foot. The parameters are sought by bringing the sole of the foot into eversion, thus bringing the scaphoid into internal rotation (the direction of correction). In order to reduce the slack, the operator drops his body weight backwards while increasing the internal rotation parameter of the scaphoid. The manipulation is performed by associating a rapid traction movement with an increase of the correction parameter towards the internal rotation of the scaphoid.
  Arms: Experimental: Osteopathic manipulation TUG for scaphoid bone
Procedure: Sham group: Sham osteopathic manipulation TUG for scaphoid bone — The intervention will be performed in the same way as the intervention group, without actually performing the TUG manipulation on the scaphoid bone, only placing it in tension.
  Arms: Sham group: Sham osteopathic manipulation TUG for scaphoid bone

SUMMARY:
This is a clinical, longitudinal, prospective and randomised study in which the subject will be assessed by stabilometric and baropodometric techniques on two occasions (before being subjected to the scaphoid tug manipulation for the experimental group or placebo technique in the case of the control group).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with right scaphoid external rotation dysfunction

Exclusion Criteria:

* Suffering from disorders that alter balance (tension headaches, vertigo, migraines...).
* Deformities, orthopaedic injuries or sequelae in the limbs or spine that may alter postural statics (valgus-varus, lower limb operations, lower limb dysmetries, scoliosis, etc.).
* Pathologies or sequelae related to the postural sensors or disorders in the same:

  * Uncorrected visual defects.
  * Vestibular disorders.
  * Uncorrected stomatological disorders.
  * Sensory alterations in the foot sensor (Hypoaesthesia, Morton's neuroma, tarsal canal syndrome, etc.).
  * Cutaneous alterations that influence the foot pick-up (papillomas, plantar warts, ingrown toenails, etc.).
  * Ingestion of medication that alters the perception of stability.
* Having any contraindication to the scaphoid tug technique.
* Having carried out intense physical activity immediately prior to the study.
* Having received osteopathic treatment in the last month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
stabilometric measurements: oscillation about the X-axis | five minutes post-intervention
  (mm)
stabilometric measurements: oscillation about the Y-axis | five minutes post-intervention
  (mm)
stabilometric measurements: area of the ellipse | five minutes post-intervention
  (cm2)
static baropodometric measurements: scan Foot bearing area | five minutes post-intervention
  (cm2)
static baropodometric measurements: scan percentage of body load supported by each foot | five minutes post-intervention
static baropodometric measurements: scan point of maximum plantar pressure | five minutes post-intervention
  (kg/cm2)

CONTACTS AND LOCATIONS:
Locations (1):
- Sergio Montero Navarro, Elche, Alicante, Spain

REFERENCES:
- [Background] Latash ML, Krishnamoorthy V, Scholz JP, Zatsiorsky VM. Postural synergies and their development. Neural Plast. 2005;12(2-3):119-30; discussion 263-72. doi: 10.1155/NP.2005.119. PMID 16097480
- [Background] Zhang Y, Kiemel T, Jeka J. The influence of sensory information on two-component coordination during quiet stance. Gait Posture. 2007 Jul;26(2):263-71. doi: 10.1016/j.gaitpost.2006.09.007. Epub 2006 Oct 13. PMID 17046262
- [Background] Myklebust JB, Prieto T, Myklebust B. Evaluation of nonlinear dynamics in postural steadiness time series. Ann Biomed Eng. 1995 Nov-Dec;23(6):711-9. doi: 10.1007/BF02584470. PMID 8572421
- [Background] Hessert MJ, Vyas M, Leach J, Hu K, Lipsitz LA, Novak V. Foot pressure distribution during walking in young and old adults. BMC Geriatr. 2005 May 19;5:8. doi: 10.1186/1471-2318-5-8. PMID 15943881
- [Background] Van Buskirk RL. Nociceptive reflexes and the somatic dysfunction: a model. J Am Osteopath Assoc. 1990 Sep;90(9):792-4, 797-809. PMID 2211195
- See also: The University CEU-Cardenal Herrera is th first private university inthe Valencian Community. It belongs to the Foundation San Pablo - CEU andis the leading educational organization in Spain with three Universities all overSpain — http://www.uchceu.es

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT05583760/Prot_SAP_ICF_000.pdf